CLINICAL TRIAL: NCT03442231
Title: Follow-Up of Subjects With a Journey™ UNI Unicompartmental Knee System Implant
Brief Title: Journey™ UNI Post Market Clinical Follow-Up
Acronym: Journey UNI
Status: Active, not recruiting | Type: Observational
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 17-4049-03
Record Dates: First submitted 2018-02-16; First posted 2018-02-22 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Non-inflammatory Degenerative Joint Disease
Keywords: osteoarthritis; traumatic arthritis; avascular necrosis
MeSH Terms: conditions — Osteoarthritis; Osteonecrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Journey™ UNI Unicompartmental Knee System: Subjects previously received knee replacement
  Interventions: Device: Journey UNI Unicompartmental Knee System

INTERVENTIONS:
Device: Journey UNI Unicompartmental Knee System — Lateral or medial knee compartment replacement

SUMMARY:
This is a retrospective/prospective, open-label single cohort, multicenter study to collect relevant clinical data from 147 subjects with unicompartmental degeneration of the knee in whom the Journey UNI UKS was previously implanted.

DETAILED DESCRIPTION:
The purpose of the current investigation is to assess the safety and effectiveness of the JOURNEY UNI Unicompartmental Knee System (UKS) in patients with non-inflammatory degenerative joint disease (NIDJD) of the knee who previously had the Journey UNI UKS implanted. This clinical study will prospectively evaluate the 36 and 60-month safety and performance of the JOURNEY UNI UKS in patients with NIDJD of the knee who required lateral or medial knee compartment replacement.

ELIGIBILITY:
Inclusion Criteria:

1. Between 12 and 48 months previously, subject had unicompartmental knee replacement implanted for unicompartmental, NIDJD including OA, traumatic arthritis, avascular necrosis, for correction of functional deformity, or to repair a fracture that was unmanageable using other techniques.
2. Subject received a Journey UKS implant (consisting of a femoral component, tibial baseplate, and a tibial insert).
3. Subject was considered skeletally mature at the time of surgery and was at least 18 years of age.
4. Subject is willing to have retrospective data collected and to participate in required prospective follow-up visit(s) at the investigational site and to complete study procedures and questionnaires.
5. Subject has consented to participate in the study by signing the Institutional Review Board (IRB)/Ethics Committee (EC)-approved informed consent form (ICF).

Exclusion Criteria:

1. Subject has Body Mass Index (BMI) > 40 within 1 month of surgery.
2. Subjects who have received the Journey UNI UKS as part of a revision surgery.
3. Subject has a condition that may interfere with the unicompartmental knee arthroplasty (UKA) survival or outcome (e.g. Paget's or Charcot's disease, vascular insufficiency, muscular atrophy, uncontrolled diabetes, moderate to severe renal insufficiency or neuromuscular disease).
4. Subject has a known allergy to study device or one or more of its components.
5. Subject, in the opinion of the Principal Investigator (PI), has an emotional or neurological condition that would preempt his/her ability or willingness to participate in the study including mental illness, mental retardation, drug or alcohol abuse.
6. Subject is entered in another investigational drug, biologic, or device study or has been treated with an investigational product in the past 30 days.
7. Subject is known to be at risk for loss to follow-up, or failure to return for scheduled visits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Investigators will pre-screen all subjects that have previously undergone UKA using the Journey UNI UKS system between 12 and 48 months previously using only the existing information in the medical records.
Sampling Method: Non-Probability Sample
Enrollment: 147 (Actual)
Dates: Start 2018-04-11 (Actual); Primary Completion 2025-04-11 (Estimated); Study Completion 2025-04-11 (Estimated)

PRIMARY OUTCOMES:
Implant survival rate | 5 years
  Did knee survive with no revision through 5 years

SECONDARY OUTCOMES:
Quality of Life - KSS | 5 Years
  2011 Knee Society Score
Quality of Life - EQ-5D - 3L | 5 Years
  EuroQol Five Dimensions Questionnaire
Quality of Life - SAPSS | 5 Years
  Self-Administered Patient Satisfaction Survey
Quality of Life - Forgotten Joint Score | 5 Years
  Forgotten Joint Score (FJS) questionnaire measures how often subject is aware of affected knee in everyday life. Score consists of 12 questions where subjects are asked to rate their awareness of their joint replacement during various activities. rating is never, almost never, seldom, sometimes or mostly.
Adverse Events (AEs) | 5 Years
  All AEs will be collected and reported
Radiographic Outcomes | 5 Years
  Perform weight-bearing AP and lateral standard x-rays

CONTACTS AND LOCATIONS:
Locations (4):
- United States (3):
  - Orthopaedic Specialists of Central Arizona-Scottsdale, Scottsdale, Arizona
  - Orthopaedic Surgery Specialists, Ltd., Park Ridge, Illinois
  - Tennesee Orthopaedic Alliance, P.A., Nashville, Tennessee
- London Health Sciences Centre-University Hospital, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No